CLINICAL TRIAL: NCT01897961
Title: Phospholipase A2 Receptor (PLA2R1) Autoantibodies in Membranous Nephropathy in Kidney Transplantation
Acronym: PRAM-KT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2011-A01302-39
Record Dates: First submitted 2012-07-20; First posted 2013-07-12 (Estimated); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Kidney Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Patients whose renal disease of origin is a GEM (Other): Patients whose renal disease of origin is a GEM
  Interventions: Other: Anticorps anti-PLA2R1
- Transplanted Patients of origin is a GEM having done it again (Other): Transplanted Patients of origin is a GEM having done it again
  Interventions: Other: Anticorps anti-PLA2R1
- Transplanted patients, and having developed a GEM of novo (Other): Transplanted patients, and having developed a GEM of novo
  Interventions: Other: Anticorps anti-PLA2R1

INTERVENTIONS:
Other: Anticorps anti-PLA2R1

SUMMARY:
The Membranous nephropathy (GEM)idiopatic is the most frequent cause of syndrome néphrotique at the adult and represent approximately 2 % of the causes of terminal chronic renal insufficiency. A etiology balance assessment must be systematically realized to eliminate a secondary cause. Antibodies managed against the receiver of phospholipases A2 secreted by type M (PLA2R1) was recently detected in a population of GEM idiopatic, but not secondary GEM. PLA2R1 is expressed by the podocytes of the glomerules of healthy subjects, and this receiver co-is located with the deposits of extramembraneous IgG of the expanding subjects of idiopathique GEM. The good IgG the extramembraneous depositsof GEM idiopathic recognize PLA2R1. At some patients, the activity anti-PLA2R1 seems to decrease or to disappear during the stake in forgiveness of the disease.

Some cases of second offense of GEM idiopathique after renal transplantation presenting antibodies anti-PLA2R1 have also described. The appearance of antibody anti-PLA2R1 seems parallel to the increase of a proteinurie in touch with a second offense of GEM, and antibodies sometimes disappeared after a therapeutic strengthening by Rituximab allowing to obtain a forgiveness.

A GEM can also appear of novo on the renal transplant, it is to say without notion of GEM on the native loins. The physiopathology of this affection remains unknown.

Working hypothesis and objectives We shall look in which proportion the presence of antibody anti-PLA2R1 is associated with the second offense of GEM idiopathic in renal transplantation. We anticipate that the GEM of novo of the renal transplant answers a different physiopathology, and will not be associated with the presence of antibody anti-PLA2R1. We hope to demonstrate that at the expanding patients of antibody anti-PLA2R1, the title of these antibodies is correlated in the activity of the disease and in the renal survival, and that the longitudinal follow-up of the title of these antibodies has an interest forecast and therapeutics.

ELIGIBILITY:
Inclusion Criteria:

* Patients of 18 or more years old,
* Presenting one of the following three profiles:
* Group 1: patients whose renal disease of origin is a GEM, and

  * or 1a: that must receive a renal transplantation, or transplanted for less than three months and having a day serum of the transplantation available on the laboratory of immunology or virology,
  * or 1b: transplanted for more than three months, not having done it again a GEM yet, and having a day serum of the transplantation available on the laboratory of immunology or virology.
* Group 2: transplanted patients whose renal disease of origin is a GEM, having done it again a GEM on their renal transplant, and having an available serum the day of the transplantation and of the diagnosis of second offense of GEM in the laboratory of immunology or virology.
* Group 3: transplanted patients, and having developed a GEM of novo, and having an available serum the day of the transplantation and of the diagnosis of GEM of novo in the laboratory of immunology or virology.

Exclusion Criteria:

* vulnerable person

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2012-01-10 (Actual); Primary Completion 2018-03-03 (Actual); Study Completion 2018-03-03 (Actual)

PRIMARY OUTCOMES:
to determine the value forecast of the presence of antibody anti-PLA2R1 | Change from baseline the presence of antibody anti-PLA2R1 at 3 month and 6 month
  to determine the value forecast of the presence of antibody anti-PLA2R1 by the reference method for the second offenseof idiopathic or secondary GEM

CONTACTS AND LOCATIONS:
Overall Officials: Vincent ESNAULT, Pr, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU de Nice, Nice, France

REFERENCES:
- [Derived] Seitz-Polski B, Dahan K, Debiec H, Rousseau A, Andreani M, Zaghrini C, Ticchioni M, Rosenthal A, Benzaken S, Bernard G, Lambeau G, Ronco P, Esnault VLM. High-Dose Rituximab and Early Remission in PLA2R1-Related Membranous Nephropathy. Clin J Am Soc Nephrol. 2019 Aug 7;14(8):1173-1182. doi: 10.2215/CJN.11791018. Epub 2019 Jul 24. PMID 31340979
- [Derived] Seitz-Polski B, Dolla G, Payre C, Tomas NM, Lochouarn M, Jeammet L, Mariat C, Krummel T, Burtey S, Courivaud C, Schlumberger W, Zorzi K, Benzaken S, Bernard G, Esnault VL, Lambeau G. Cross-reactivity of anti-PLA2R1 autoantibodies to rabbit and mouse PLA2R1 antigens and development of two novel ELISAs with different diagnostic performances in idiopathic membranous nephropathy. Biochimie. 2015 Nov;118:104-15. doi: 10.1016/j.biochi.2015.08.007. Epub 2015 Aug 19. PMID 26296473